CLINICAL TRIAL: NCT07246135
Title: Leadless Pacemaker Registry
Brief Title: Leadless Pacemaker Registry: Outcomes and Follow-up From the University Hospital of St. Pölten
Acronym: LPR
Status: Recruiting | Type: Observational
Sponsor: Karl Landsteiner University of Health Sciences (Other)
Collaborators: University Hospital St. Polten (Other)
Responsible Party: Sponsor
Other Study IDs: GS3-EK-4/899-2024
Record Dates: First submitted 2025-09-16; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-09

CONDITIONS: Pacemaker; Leadless Pacemaker; Cardiac Pacing, Artificial; Registries
Keywords: Registry; Leadless Pacemaker; Pacemaker; Cardiac Pacing; Pacemaker Complication; Leadless Pacemaker Outcomes; Heart Conduction System Disease; Bradycardia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The registry for leadless pacemakers will collect and annually analyze the data of all leadless pacemaker implantations at the University Hospital St. Pölten, including demographic information, indications, procedural details, acute, medium- and long-term complications during follow-up. Due to the partially novel nature of the signals (atrial mechanical sensing markers) and the lack of long-term experience to date, data on these aspects will also be collected and analyzed.

This is a single-center, prospective and retrospective registry that includes all patients receiving a leadless pacing device, as well as all patients who received a leadless pacing device between January 2021 and the start of the registry. All patients undergoing implantation of a leadless pacemaker will be invited to participate in the registry. For patients to be included retrospectively, participation in the registry will be offered at the time of their next routine follow-up visit.

The indication for leadless pacing will be determined by the physician responsible for the patient. Enrollment in the registry will in no case alter or influence the treatment the patient receives. Data collection will take place at the time of implantation and continuously during follow-up over the entire study period. Pacemaker-related data may be obtained either in person or via remote monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing implantation of a leadless pacemaker at the University Hospital of St. Pölten
* Patients who previously received a leadless pacemaker between June 2015 and the start of the registry (retrospective inclusion).
* Age ≥ 18 years.
* Written informed consent provided by the patient.

Exclusion Criteria:

* Patients who decline or are unable to provide informed consent.
* Patients in whom a conventional transvenous pacemaker is implanted (i.e., not leadless).
* Any condition that, in the opinion of the treating physician, precludes participation in the registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients undergoing implantation of a leadless pacemaker at University Hospital St. Pölten, as well as patients who previously received a leadless pacemaker at the same institution since June 2015. Both prospective and retrospective patients are included.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2015-06-18 (Actual); Primary Completion 2035-01 (Estimated); Study Completion 2035-01 (Estimated)

PRIMARY OUTCOMES:
Procedural success rate | Periprocedural / at Day 1
  Successful implantation of a leadless pacemaker with acceptable electrical parameters and no need for conversion to a transvenous system
Incidence of acute complications | Within 30 days after implantation
  Rate of periprocedural complications (e.g., vascular complications, arrhythmias, pericardial effusion, device dislodgement)

SECONDARY OUTCOMES:
Device-related complication rate (medium- and long-term) | Up to 10 years after implantation
  Cumulative incidence of complications requiring medical or surgical intervention (e.g., device malfunction, infection, need for extraction, upgrade)
Ventricular pacing burden | Day 1, 3 months post-implant (±2 weeks), 1 year after Implantation (±2 weeks), every 12th month (±2 weeks) thereafter
  Percentage of ventricular pacing and triggered pacing as recorded by device interrogation
All-cause mortality | Throughout follow-up (up to 10 years)
Hospitalizations related to cardiac arrhythmias or heart failure | Throughout follow-up (up to 10 years)
Quality of Life after Implantation | 1 year after Implantation (±2 weeks), every 12th month (±2 weeks) thereafter
  Change in 12-Item Short Form Health Survey (SF-12) questionnaire score / The SF-12 questionnaire is a validated health-related quality of life instrument with two subscales: Physical Component Summary (PCS) and Mental Component Summary (MCS). Each subscale ranges from 0 to 100 points, where higher scores indicate better health-related quality of life.
Electrical performance of the device | Day 1, 3 months post-implant (±2 weeks), 1 year after Implantation (±2 weeks), every 12th month (±2 weeks) thereafter
  Pacing thresholds (in Volts at 0.24 ms pulse width)
Electrical performance of the device | Day 1, 3 months post-implant (±2 weeks), 1 year after Implantation (±2 weeks), every 12th month (±2 weeks) thereafter
  Sensing Amplitude (R-wave, in millivolts [mV])
Electrical performance of the device | Day 1, 3 months post-implant (±2 weeks), 1 year after Implantation (±2 weeks), every 12th month (±2 weeks) thereafter
  Lead impedance (in Ohms [Ω])
Electrical performance of the device | Day 1, 3 months post-implant (±2 weeks), 1 year after Implantation (±2 weeks), every 12th month (±2 weeks) thereafter
  Estimated battery longevity (in years)
Left ventricular ejection fraction on Echocardiography | 1 year after Implantation (±2 weeks), every 12th month (±2 weeks) thereafter
  in %
Left ventricular dimensions on Echocardiography | 1 year after Implantation (±2 weeks), every 12th month (±2 weeks) thereafter
  end-diastolic and end-systolic diameters, in mm
Right ventricular function on Echocardiography | 1 year after Implantation (±2 weeks), every 12th month (±2 weeks) thereafter
  Tricuspid Annular Plane Systolic Excursion (TAPSE) in mm

CONTACTS AND LOCATIONS:
Overall Officials: Julia Mascherbauer, MD, Professor, Principal Investigator — Department of Internal Medicine III, University Hospital of St. Pölten
Locations (1):
- University Hospital of St. Pölten, Sankt Pölten, Lower Austria, Austria

IPD SHARING:
Plan to Share IPD: No